CLINICAL TRIAL: NCT01534312
Title: Casein Glycomacropeptide in Active Distal Ulcerative Colitis (Pilot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Arla Foods (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGMP in UC
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2012-12

CONDITIONS: Colitis, Ulcerative; Inflammatory Bowel Diseases
Keywords: Glycopeptides; Dietary proteins
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CGMP protein (Experimental): Casein glycomacropeptide 30 gram/day, unchanged prophylactic 5ASA dose
  Interventions: Drug: CGMP protein
- Standard oral 5ASA maximal dose (Active Comparator): Increase from prophylactic dose 5ASA (mesalazine) to maximal oral dose, i.e. 4800 grams of mesalazine (Asacol/Mezavant)
  Interventions: Drug: Maximal oral 5ASA

INTERVENTIONS:
Drug: CGMP protein — Casein glycomacropeptide purified powder dissolved in 300 ML water once daily
  Other Names: Casein glycomacropeptide
  Arms: CGMP protein
Drug: Maximal oral 5ASA — 4800 grams/day of Mesalazine (Asacol/Mezavant)
  Other Names: Asacol; Mezavant; Mesalazine
  Arms: Standard oral 5ASA maximal dose

SUMMARY:
Casein glycomacropeptide (CGMP) has anti-inflammatory properties in experimental rodent colitis and using human in vitro inflammation models. Its use as a food ingredient has proven safe and with no influence on dietary intake. We hypothesize that orally administered CGMP has a beneficial effect comparable to that of mesalazine in active distal ulcerative colitis.

DETAILED DESCRIPTION:
GCMP has mainly been used as food additive in patients with specific dietary needs, i.e. in infant formulas, adipositas, or in patient with phenylketonuria. Due to its antiinflammatory properties we hypothesize that it may be used alone or along with conventional therapy in inflammatory diseases such as ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* Diagnosed ulcerative colitis
* Signs of clinical activity with SCCAI of 3 or more
* Extension more than 10 cm and no more than 40 cm from anus

Exclusion Criteria:

* Rectal temperature more than 38 degrees Celcius
* Diagnosed celiac disease or lactose intolerance
* Unable to speak or understand Danish
* Prior biologics or systemic steroids 4 weeks up to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Fecal calprotectin reduction | 4 weeks
  Relative reduction in fecal calprotectin measured before and after 4 weeks

SECONDARY OUTCOMES:
Clinical activity index | 4 weeks
  Simple Clinical Colitis Index, range 0-20
Quality of life | 4 weeks
  Quality of life measured yb Short Health Scale (4 items ranged 0-10, total range 0-40)
Endoscopic Mayo score | 4 weeks
  Grade of inflammation (range 0-3) in rectum according to Mayo score, visually judged during endoscopy
Serial fecal calprotectin | 8 weeks
  fecal calprotectin week 0-4-6-8

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Vilstrup, Professor, Study Chair — Professor, University of Aarhus
Locations (1):
- Department of medicine V (Hepatology and Gastroenterology), Aarhus C, Aarhus C, Denmark